CLINICAL TRIAL: NCT00903019
Title: Telehealth Problem-Solving Therapy for Depressed Homebound Older Adults
Brief Title: Feasibility of Telehealth Problem-Solving Therapy for Depressed Homebound Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Namkee Choi, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R34MH083872 (NIH); R34MH083872 (NIH); DATR A4-GPS
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Depression
Keywords: Homebound; Older Adults; Disability; Videoconferencing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive problem-solving therapy (PST) delivered via teleconferencing (tele-PST).
  Interventions: Behavioral: Tele-Problem-Solving Therapy
- 2 (Active Comparator): Participants will receive problem-solving therapy (PST) delivered in-person.
  Interventions: Behavioral: In-Person PST
- 3 (Placebo Comparator): Participants will receive monitoring phone calls.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Tele-Problem-Solving Therapy — Six sessions of tele-PST
  Arms: 1
Behavioral: In-Person PST — Six sessions of in person PST
  Arms: 2
Behavioral: Attention control — Six weekly telephone calls
  Arms: 3

SUMMARY:
This study will test the feasibility and effectiveness of therapy given via teleconferencing to depressed homebound older adults.

DETAILED DESCRIPTION:
Older people with disabilities who cannot leave their homes are at increased risk of depression or depressive symptoms. Short-term psychotherapy, without medications, has been found effective for treating this population of people. Problem-solving therapy (PST) is a brief, structured, cognitive-behavioral therapy that teaches people problem-solving and coping skills to deal with negative life events and daily problems. Previous research demonstrated that PST is an effective treatment for depression when delivered to older adults in their homes. The cost of service for these in-home visits, however, can be prohibitive for many older adults and social service providers. One way to extend treatment to more older adults is to deliver PST via teleconferencing (tele-PST). This study will test the feasibility and effectiveness of tele-PST in treating depression in homebound older adults.

This study will have two phases. Phase 1 will examine the feasibility of delivering treatment via teleconference. Participants in this phase will receive six weekly sessions of tele-PST and then complete a 2-week follow-up visit in which their depression, disability, and resourcefulness will be assessed. Logistical and procedural problems and acceptability of the treatment to participants will be used to guide modifications or adaptations made to tele-PST before conducting a larger, randomized trial in Phase 2.

Participation in Phase 2 will last 6 weeks, with follow-up visits lasting until 24 weeks after the conclusion of treatment. Participants will be randomly assigned to one of three groups: tele-PST, in-person PST, and attention control. Participants in the tele-PST group will receive six weekly sessions of PST via teleconference, and participants in the in-person PST group will receive six weekly sessions of PST from a study therapist in person. Both these groups will also receive six monthly maintenance calls from their study therapist after the completion of treatment. Participants in the attention group will receive six weekly phone calls followed by six monthly phone calls to monitor their health. All participants in Phase 2 will complete assessments at 2, 12, and 24 weeks following their treatment. These assessments will measure the adequacy of recruitment, enrollment, and retention strategies; the compliance rates and service delivery costs of tele-PST and in-person PST; and participants' depression, disability, and resourcefulness.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic white, African American, or Hispanic
* Homebound, as defined by receiving a home-delivered meals service or personal assistance and in-home support services because of disability
* Moderate-to-severe depressive symptom severity, as defined by a score greater than or equal to 15 on the Hamilton Rating Scale for Depression (HAMD)
* Has a home television set that can be used for problem-solving therapy (PST) sessions
* Has a landline telephone

Exclusion Criteria:

* High suicide risk, as defined by an intent or plan to attempt suicide within a month or indication of persistently moderate or severe suicidal ideation or behavior
* Presence of dementia or executive dysfunction
* Presence of bipolar disorder
* Lifetime or current (within 12 months) psychotic symptoms or disorder
* Presence of co-occurring alcohol or other addictive substance abuse, including benzodiazepines and opioids
* Hearing or vision impairment that would interfere with PST participation
* Inability to actively participate in PST sessions due to acute or severe medical illness or functional impairment, such as a bed-bound state
* Current involvement in psychotherapy
* Inability to speak English

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
24-item Hamilton Rating Scale for Depression (HAMD) | Measured at 2, 12, and 24 weeks
12-item World Health Organization Disability Assessment Schedule (WHO-DAS-II) | Measured at 2, 12, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Namkee G. Choi, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Choi NG, Marti CN, Bruce ML, Kunik ME. Relationship between depressive symptom severity and emergency department use among low-income, depressed homebound older adults aged 50 years and older. BMC Psychiatry. 2012 Dec 26;12:233. doi: 10.1186/1471-244X-12-233. PMID 23267529